CLINICAL TRIAL: NCT07275775
Title: A Phase I, Randomized, Double-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose and Food Effect Study to Evaluate the Safety, Tolerability and Pharmacokinetics of D-2570 Tablets in Healthy Subjects
Brief Title: Single and Multiple Dose and Food Effect Study to Evaluate the Safety, Tolerability and Pharmacokinetics of D-2570 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D2570-102
Record Dates: First submitted 2024-11-04; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Compare the safety and tolerability of D-2570 tablets with Placebo for evaluation (Experimental): To assess the safety and tolerability of single, multiple doses and food effect trial of D-2570 tablets and Placebo in healthy subjects.
  Interventions: Drug: D-2570; Drug: Placebo
- Characterize the pharmacokinetics of single, multiple doses of D-2570 tablets and Placebo (Experimental): To characterize the pharmacokinetics (PK) of single, multiple doses of D-2570 tablets and Placebo in healthy subjects.
  Interventions: Drug: D-2570; Drug: Placebo
- Compare the effects of D-2570 with Placebo on the QT/QTc interval for assess (Experimental): To assess the effects of D-2570 and Placebo on the QT/QTc interval in healthy subjects.
  Interventions: Drug: D-2570; Drug: Placebo
- Compare the effects of multiple doses D-2570 with Placebo on serum IL-17A (Experimental): To assess the effects of multiple doses D-2570 and Placebo on serum IL-17A in healthy subjects.
  Interventions: Drug: D-2570; Drug: Placebo
- Assess the effects of regular and high-fat on the pharmacokinetics of D-2570 tablets (Experimental): To assess the effects of regular and high-fat on the pharmacokinetics of D-2570 tablets.
  Interventions: Drug: D-2570
- Evaluate the relative bioavailability among health benefits of D-2570 tablets (9 mg specification) (Experimental): To evaluate the relative bioavailability among health benefits of D-2570 tablets (9 mg specification) and D-2570 tablets (3 mg specification)
  Interventions: Drug: D-2570

INTERVENTIONS:
Drug: D-2570 — D-2570 is a novel inhibitor targeting the TYK2 pseudokinase domain, which can inhibit the release of inflammatory factors and participate in immune regulation. D-2570 is being developed as a potential oral therapeutic drug for patients with psoriasis, ulcerative colitis, SLE, and other conditions.
Drug: Placebo — A placebo refers to a tablet that has no therapeutic effect on medication.
  Arms: Characterize the pharmacokinetics of single, multiple doses of D-2570 tablets and Placebo; Compare the effects of D-2570 with Placebo on the QT/QTc interval for assess; Compare the effects of multiple doses D-2570 with Placebo on serum IL-17A; Compare the safety and tolerability of D-2570 tablets with Placebo for evaluation

SUMMARY:
This is a randomized, double-blind, placebo-controlled single and multiple ascending dose and food effect study on PK. Subjects in the SAD and MAD study take the drug under fasting conditions, while those in the food effect (FE) study are required to take the drug under fasting or fed conditions according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily take part in the study after being fully informed, sign a written informed consent form (ICF), and agree to follow procedures specified in the study protocol;
* Subjects who can take effective contraceptive measures from the start of screening to 6 months after the last dose of the IMP;
* Male and female subjects aged 18 to 45 years (inclusive);
* Male weight ≥ 50 kg, female weight ≥ 45 kg. Body mass index (BMI) = body weight (kg) / height2 (m2). BMI ranging from 19 to 26 kg/m2 (inclusive);
* Subjects without medical history of clinically significant respiratory, circulatory, digestive, urinary, hematological, endocrine, nervous system diseases, metabolic abnormalities or infections, etc.

Exclusion Criteria:

* More than 5 cigarettes per day on average within 3 months before screening;
* Subjects with a clinically significant history of drug allergy or specific allergic diseases (asthma, urticaria) or known allergy to the IMP or its excipients;
* History of alcohol abuse (consuming an average of 14 units of alcohol per week within 3 months prior to screening: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
* Subjects with a history of substance or drug abuse or a positive urine drug screening;
* Blood donation or massive blood loss (>450 mL) within 3 months before screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | During the procedure
  Incidence of adverse events
Result of vital signs | During the procedure
  Test of resting blood pressure.
Result of vital signs | During the procedure
  Test of resting heart pulse.
Result of vital signs | During the procedure
  Test of respiratory rate.
Result of vital signs | During the procedure
  Test of body temperature.
Result of physical examination | During the procedure
  Test of height (meters）
Result of physical examination | During the procedure
  Test of weight (kilograms)
Result of electrocardiogram | During the procedure
  Test of beats per minute
Result of electrocardiogram | During the procedure
  Test of RR Interva
Result of electrocardiogram | During the procedure
  Test of PR Interva
Result of electrocardiogram | During the procedure
  Test of QRS Interva
Result of electrocardiogram | During the procedure
  Test of QT Interva
Result of electrocardiogram | During the procedure
  Test of QTcF msec
Result of PK endpoints | Day1 to Day7 of group SAD
  Tmax
Result of PK endpoints | Day1 to Day13 of group MAD
  Tmax
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  Tmax
Result of PK endpoints | Day1 to Day7 of group SAD
  Cmax
Result of PK endpoints | Day1 to Day13 of group MAD
  Cmax
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  Cmax
Result of PK endpoints | Day1 to Day7 of group SAD
  t1/2
Result of PK endpoints | Day1 to Day13 of group MAD
  t1/2
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  t1/2
Result of PK endpoints | Day1 to Day7 of group SAD
  MRT
Result of PK endpoints | Day1 to Day13 of group MAD
  MRT
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  MRT
Result of PK endpoints | Day1 to Day7 of group SAD
  AUC0-∞
Result of PK endpoints | Day1 to Day13 of group MAD
  AUC0-∞
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  AUC0-∞
Result of PK endpoints | Day1 to Day7 of group SAD
  AUC0-t
Result of PK endpoints | Day1 to Day13 of group MAD
  AUC0-t
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  AUC0-t
Result of PK endpoints | Day1 to Day7 of group SAD
  CL/F
Result of PK endpoints | Day1 to Day13 of group MAD
  CL/F
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  CL/F
Result of PK endpoints | Day1 to Day7 of group SAD
  Vz/F
Result of PK endpoints | Day1 to Day13 of group MAD
  Vz/F
Result of PK endpoints | Day1 to Day7 for every cycle of group FE
  Vz/F
Assessment of hematology test | During the procedure
  Red blood cell count
Assessment of hematology test | During the procedure
  Hemoglobin measurement
Assessment of hematology test | During the procedure
  Hematocrit measurement
Assessment of hematology test | During the procedure
  Platelet count
Assessment of hematology test | During the procedure
  White blood cell count
Assessment of hematology test | During the procedure
  Lymphocyte count
Assessment of hematology test | During the procedure
  Neutrophil count
Assessment of hematology test | During the procedure
  Monocyte count
Assessment of hematology test | During the procedure
  Eosinophil count
Assessment of hematology test | During the procedure
  Basophil count
Assessment of urinalysis test | During the procedure
  pH measurement
Assessment of urinalysis test | During the procedure
  Protein detection
Assessment of urinalysis test | During the procedure
  White blood cells count
Assessment of urinalysis test | During the procedure
  Red blood cells count
Assessment of urinalysis test | During the procedure
  Glucose measurement
Assessment of urinalysis test | During the procedure
  Specific gravity measurement
Assessment of coagulation parameters test | During the procedure
  Thrombin time
Assessment of coagulation parameters test | During the procedure
  Partial thromboplastin time
Assessment of coagulation parameters test | During the procedure
  International normalized ratio
Assessment of coagulation parameters test | During the procedure
  Fibrinogen
Assessment of blood biochemistry test | During the procedure
  Sodium
Assessment of blood biochemistry test | During the procedure
  Potassium
Assessment of blood biochemistry test | During the procedure
  Calcium
Assessment of blood biochemistry test | During the procedure
  Chlorine
Assessment of blood biochemistry test | During the procedure
  Total protein
Assessment of blood biochemistry test | During the procedure
  Albumin
Assessment of blood biochemistry test | During the procedure
  Alkaline phosphatase
Assessment of blood biochemistry test | During the procedure
  Alanine aminotransferase
Assessment of blood biochemistry test | During the procedure
  Aspartate aminotransferase
Assessment of blood biochemistry test | During the procedure
  Direct bilirubin
Assessment of blood biochemistry test | During the procedure
  Indirect bilirubin
Assessment of blood biochemistry test | During the procedure
  Total bilirubin
Assessment of blood biochemistry test | During the procedure
  Gamma glutamyl transferase
Assessment of blood biochemistry test | During the procedure
  Uric acid
Assessment of blood biochemistry test | During the procedure
  Creatinine
Assessment of blood biochemistry test | During the procedure
  Creatine kinase
Assessment of blood biochemistry test | During the procedure
  Urea
Assessment of blood biochemistry test | During the procedure
  Glucose
Assessment of blood biochemistry test | During the procedure
  Total cholesterol
Assessment of blood biochemistry test | During the procedure
  Triglycerides

SECONDARY OUTCOMES:
Result of safety endpoint | During the procedure
  Test of QT Interva.
Result of safety endpoint | During the procedure
  Test of QTc Interva.
Result of PD endpoint | Day1 of group SAD
  Test of serum IL-17A.
Result of PD endpoint | Day1 and Day7 of group MAD
  Test of serum IL-17A.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuguang Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No